CLINICAL TRIAL: NCT00180349
Title: Short and Long Term Evaluation of Electrical Measurements and Defibrillation Energies, Results of ATP and Diagnostic Functions of Devices Connected to Endotak RELIANCE® Defibrillation Leads
Brief Title: Leader - Evaluation of Endotak Reliance
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Leader v. 1.0 10/04
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Endotak Reliance — Endotak Reliance is a defibrillation lead delivering pacing and defibrillation therapy to the ventricle as needed.

SUMMARY:
The objective of this study is to demonstrate the efficacy of the ENDOTAK® RELIANCE™ defibrillation leads connected to a defibrillator or a cardiac resynchronization defibrillator from implant until 12 months.

DETAILED DESCRIPTION:
Baseline and clinical data were collected at inclusion, as were data on procedural characteristics, device implantation-related adverse events and device programming at the time of hospital discharge. Patients were subsequently divided in two groups: patients who underwent VF induction at implantation or before hospital discharge(VF induction group); and patients who did not undergo VF induction (untested group).The patients were followed up at 3-6 months and at12 months after the implantation. VF induction procedures were left to the investigator's discretion, but reasons for not performing a VF induction at implantation were recorded prospectively. ICD programming parameters for tachycardia or bradycardia were also left at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* ICD indication according to current guidelines with or without cardiac resynchronization therapy, being implanted with a Guidant ENDOTAK RELIANCE defibrillation lead as first implant, age above 18 years, able to understand the nature of the study and to be available for all follow-ups, having given consent in writing for anonymous data collection, life expectancy > 1 year.

Exclusion Criteria:

* device replacement without concomitant implant of a Reliance defibrillation lead, pregnancy or of birth bearing age without contraception, participation in another clinical study, short life expectancy due to other medical conditions, not willing to sign the consent form, geographically unstable for a defibrillator follow-up as required per protocol, having a ventricular arrhythmia, that can be treated by drugs or surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with the indication for an implantable ICD are invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 904 (Actual)
Dates: Start 2004-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Defibrillation testing (DT) procedures and consequences on clinical outcomes | at implant
  to determine the DT procedures used in everyday practice, to compare the characteristics of patients with or without DTand to compare severe adverse events in these two populations during implantation
Defibrillation testing (DT) procedures and consequences on clinical outcomes | during 1 year follow-up
  to determine the DT procedures used in everyday practice, to compare the characteristics of patients with or without DTand to compare severe adverse events in these two populations during 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Sadoul, MD, Principal Investigator — CHU Brabois, Nancy; Arnaud Lazarus, MD, Principal Investigator — Clinique Bizet, Paris
Locations (25):
- France (25):
  - CH Amiens, Amiens
  - CHU Angers, Angers
  - Hôpital Angoulème, Angoulème
  - Clinique Cardiologique Aressy, Aressy
  - CH Avignon, Avignon
  - CHU du Morvan, Brest
  - Hôpital Côte de Nacre, Caen
  - CHU Henri Mondor, Créteil
  - CHU Michalon, Grenoble
  - CH Hôpital Nord, Marseille
  - CHU La Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHU Brabois, Nancy
  - Nouvelle Clinique Nantaise, Nantes
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - CHU D'Orleans, Orléans
  - Clinique Bizet, Paris
  - CHG Pau, Pau
  - CHU Pontchaillou, Rennes
  - CHU Rouen, Rouen
  - Centre cardiologique du Nord, Saint-Denis
  - CMC Arnaud Tzanck, Saint-Laurent-du-Var
  - CHU Rangueil, Toulouse
  - Clinique St. Gatien, Tours